CLINICAL TRIAL: NCT04864132
Title: The Investigation Of Exercise Capacity And Exercise-Induced Fatigue in Young Adults Who Survived From Coronavirus
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Associated Proffesor, Biruni University
Other Study IDs: 2015-KAEK-47-21-03
Record Dates: First submitted 2021-04-20; First posted 2021-04-28 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: coronavirus; exercise capacity
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Walk Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects survived from COVID-19: The subjects who had confirmed COVID-19 infection aged between 18-30/years
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: Incremental shuttle walk test
- Subjects never had COVID-19: The subjects aged between 18-30/years who have not been diagnosed with COVID-19 as of March 11of 2020 and who have not been in contact and risky according to the "Life Fits Into Home" application
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: Incremental shuttle walk test

INTERVENTIONS:
Diagnostic Test: 6-minute walk test — This test assesses submaximal exercise capacity.
Diagnostic Test: Incremental shuttle walk test — This test assesses maximal exercise capacity.

SUMMARY:
The effects of Coronavirus Disease (COVID-19), a multisystem disease, on the body system and functions are being investigated all over the world. Examining the effect of exercise capacity, which is an important marker of cardiovascular risk in young individuals with COVID-19, will allow the planning of exercise and physical activity programs according to the needs of that specific population. The objectives of this project are:(1) To compare the submaximal and maximal exercise capacity of young adults aged between 18-30 who have had COVID-19 with healthy individuals in the same age group (2) To determine the roles of muscle strength, respiratory functions, fatigue, dyspnea, and physical activity level on exercise capacity evaluated by two different tests in young adults survived from COVID-19.

DETAILED DESCRIPTION:
The effects of COVID-19, a multisystem disease, on the body system and functions are being investigated worldwide. For young adults, exercise capacity is vital in the workforce, cardiovascular risk factors and long-term health perception. Determining exercise capacity, which is an essential indicator of cardiovascular risk in the long term, and determining the factors affecting exercise capacity in cases with COVID-19 will allow the planning of exercise and physical activity programs according to young people's needs. The objectives of this project are:(1) To compare the submaximal and maximal exercise capacity of young adults aged between 18-30 who have had COVID-19 with healthy individuals in the same age group (2) To determine the roles of muscle strength, respiratory functions, fatigue, dyspnea, and physical activity level on exercise capacity evaluated by two different tests in young adults survived from COVID-19. There is no study in the literature evaluating the exercise capacity and the factors affecting the prolonged COVID-19 symptoms for patients with COVID-19. This project can provide objective evidence on this subject and includes controlled multi-directional measurement.

ELIGIBILITY:
Inclusion Criteria:

* For cases with COVID-19:

Confirmed COVID-19 infection - For healthy individuals of the same age group who have not had COVID-19: Individuals who have not been diagnosed with COVID-19 as of March 11, 2020 and who have not been in contact and risky according to the "Life Fits Into Home" application

- For all participants; Answering "No" to all questions in the Physical Activity Readiness Questionnaire.

Exclusion Criteria:

* Individuals with orthopedic or neurological disabilities that may interfere with exercise testing,
* Individuals with a fever> 38 ° C and / or resting blood pressure <90/60 mmHg or> 140/90 mmHg and/or oxygen saturation ≤95%,
* Individuals who have been involved in a physiotherapy and rehabilitation program within the last 3 months,
* Individuals with insufficient cooperation
* Individuals with blood coagulation disorders contraindicated for blood lactate analysis,
* Pregnant women or individuals with suspected pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects who survived from COVID-19 aged between 18-30 and healthy individuals in the same age will be included in the project.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Submaximal and maximal exercise tests | 1 year
  The 6 minutes walking distance and incremental shuttle walk distance will be measured.

SECONDARY OUTCOMES:
Fatigue Severity Scale | 1 year
  Fatigue levels will be measured with this scale. This questionnaire contains nine statements that rate the severity of your fatigue symptoms and each question ranged from 1 to 7 based on how accurately it reflects the condition of the participant during the past week.
Dyspnea-12 Scale | 1 year
  The dyspnea perception will be measured with this scale.There are 12 descriptor items on this scale ranging none (0), mild (1), moderate (2), or severe (3). It provides an overall score for breathlessness severity that incorporates seven physical items and five affective items.
International Physical Activity Questionnaire-Short Form (IPAQ) | 1 year
  The physical activity (PA) levels will be measured with this scale.The IPAQ-short is a seven-item measure of vigorous-intensity physical activity, moderate-intensity physical activity, walking, and sitting. Participants reported physical activity frequency, duration, and total time spent sitting on a week day during the last week. The total daily PA (MET-min day21) will be estimated by summing the multiplication of reported time within each item by a MET value specific to each category of PA and expressed as a daily average MET score, in accordance with the official IPAQ scoring protocol.
Forced expiratory volume in first second (FEV1) (predicted %) | 1 year
  The acceptance criteria of the American Thoracic Society/European Respiratory Society will be used for spirometric measurements.
Peripheral muscle strength | 1 year
  The upper and lower extremity muscle strength will be measured using hand held dynamometer.
Respiratory muscle strength | 1 year
  Maximal inspiratory (MIP) and expiratory pressures (MEP) will be measured. Maximal inspiratory pressure will be assessed from the residual volume and MEP will assessed a using the total lung capacity.
Forced vital capacity (FVC) (predicted %) | 1 year
  The acceptance criteria of the American Thoracic Society/European Respiratory Society will be used for spirometric measurements.
FEV1/FVC (predicted %) | 1 year
  The acceptance criteria of the American Thoracic Society/European Respiratory Society will be used for spirometric measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akinci, Assoc. Prof., Study Chair — Biruni University; Zeynep Hosbay, Assoc. Prof., Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)